CLINICAL TRIAL: NCT04043351
Title: Diagnostic Performance of Exome Sequencing in Autism Spectrum Disorders
Acronym: REDIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/0417/HP
Record Dates: First submitted 2019-07-23; First posted 2019-08-02 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluation of the diagnostic performance of exome sequencing in a prospective series of patients with autism spectrum disorders (ASD).

ELIGIBILITY:
Inclusion Criteria:

* Patient with ASD who has been previously diagnosed by an expert center according to the DSM5 criteria using standardized instruments (ADOS, ADI-R), referred to genetic consultation by the psychiatrist who performed the clinical diagnosis, according to the recommendations of the HAS, and requesting a genetic analysis for medical purposes in this context.
* Patient over 3 years old
* Patient affiliated to a social security scheme
* For minor patients: Holders of the exercise of parental authority who have read and understood the newsletter and signed the consent form
* For a major patient: Major patient who has read and understood the newsletter and signed the consent form
* Supervised minor / minor patient: Legal representative who has read and understood the newsletter and signed the consent form
* Major patient under guardianship: Major patient assisted by his curator or by the judge having read and understood the newsletter and signed the consent form
* DNA of the patient and parents available

Exclusion Criteria:

* Patient who has already benefited from exome sequencing
* Person deprived of liberty by an administrative or judicial decision
* Pregnant or lactating woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Autism Spectrum Disorder (ASD)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Proportion of unrelated index cases | through study completion, an average of 4 years
  at least one definite or probable risk factor or causal variant of a monogenic form of autism

CONTACTS AND LOCATIONS:
Overall Officials: GAEL NICOLAS, Principal Investigator — ROUEN HOSPITAL
Locations (1):
- DRCI, Rouen, France